CLINICAL TRIAL: NCT05838092
Title: A Double-blind, Randomized, Placebo-controlled, Interventional, Multicenter, Phase III Clinical Trial to Investigate the Safety and Efficacy of ABCB5-positive Mesenchymal Stromal Cells (ABCB5+ MSCs) on Epidermolysis Bullosa (EB)
Brief Title: Allogeneic ABCB5-positive Dermal Mesenchymal Stromal Cells for Treatment of Epidermolysis Bullosa (Phase III)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: allo-APZ2-EB-III-01
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental)
  Interventions: Drug: allo-APZ2-OTS
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: allo-APZ2-OTS — Allogeneic dermal ABCB5-positive Mesenchymal Stromal Cells (ABCB5+ MSCs)
  Arms: Verum
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to investigate the safety and efficacy of allo-APZ2-OTS administered intravenously to subjects with recessive dystrophic epidermolysis bullosa (RDEB) compared to placebo. An additional baseline-controlled open-label arm will be included to investigate the safety and efficacy of allo-APZ2-OTS administered intravenously to subjects with JEB and to RDEB subjects < 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects from 6 months of age with a diagnosis of RDEB confirmed by genetic testing or by a skin biopsy with immunofluorescence mapping
2. Subject is eligible to participate in this clinical trial based on general health condition;
3. Subject with a target wound meeting the following criteria: 5-50 cm2, ≥ 21 days and < 9 months, no signs of acute infection;
4. Patient/legal representative understands the nature of the procedure and provide written informed consent/assent prior to any clinical trial procedure;
5. Women of childbearing potential must have a negative urine pregnancy test at Visit 1. Women of childbearing potential, male participants, and their partner must be willing to use highly effective contraceptive methods during the course of the entire clinical trial.

Exclusion Criteria:

1. Any current tumor diseases, including squamous cell carcinoma and basal cell carcinoma;
2. Any known allergies to components of the IP or premedication;
3. Patient/legal representative anticipated to be unwilling or unable to comply with the requirements of the protocol;
4. Pregnant or lactating women;
5. Current or previous (within 30 days of screening) treatment with another IP, or participation and/or under follow-up in another interventional clinical trial;
6. Previous participation in this clinical trial (except for screening failures);
7. Clinically significant or unstable concurrent disease or other clinical contraindications like an uncontrolled or poorly controlled mental health condition of the subject and/or his/her legal representative that could impact on patient's safety or interfere with study compliance such as inability to attend scheduled study visits; Confidential
8. Employees of the sponsor, or employees or relatives of the investigator.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with complete target wound closure | 6 Months
  Proportion of subjects with complete healing of target wound, determined by the investigator, as compared to baseline

SECONDARY OUTCOMES:
Time to complete target wound closure from baseline | 6 Months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Masonic Cancer Center and Medical Center Minneapolis, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided